CLINICAL TRIAL: NCT02708329
Title: Results of T-provisional and Mini Crush Stenting in Patients With Bifurcation Lesions After Chronic Coronary Arteries Occlusions Recanalization: A Prospective Randomized Single-center Study.
Brief Title: T-provisional Stenting vs Mini-Crush in Chronic Total Occlusions (CTO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TvsMC 1.0
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Ischemic Heart Disease; Coronary Atherosclerosis; Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Coronary stenosis; Drug-eluting stent; Coronary angioplasty with stenting; Ischemic Heart Disease; Chronic total occlusion; Bifurcational lesion; Bifurcational stenting
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Coronary Stenosis

ARMS (2):
- CTO coronary angioplasty +T-provisional stenting (Active Comparator): Coronary angioplasty using T-provisional stenting in patients with bifurcational lesion in Chronic total occlusion segment.
  Interventions: Procedure: T-provisional stenting; Procedure: CTO coronary angioplasty
- CTO coronary angioplasty + Mini-crush stenting (Experimental): Coronary angioplasty using Mini-crush stenting in patients with bifurcational lesion in Chronic total occlusion segment.
  Interventions: Procedure: Mini-crush stenting; Procedure: CTO coronary angioplasty

INTERVENTIONS:
Procedure: T-provisional stenting — Standard endovascular T-provisional stenting technique
  Arms: CTO coronary angioplasty +T-provisional stenting
Procedure: Mini-crush stenting — Standard endovascular Mini-crush stenting technique
  Arms: CTO coronary angioplasty + Mini-crush stenting
Procedure: CTO coronary angioplasty — A standard endovascular procedure is carried out under local anesthesia and under fluoroscopic control. Recanalisation of coronary artery CTO is performed by the hydrophilic coronary wire, using the most appropriate technique. Then balloon angioplasty of target lesion is provided. After the angiographic control coronary stent is implanted. After coronary wire removing control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix(clopidogrel) in dose 300-600 mg prescription before the procedure and heparin (heparin sodium) injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix(clopidogrel) in dose 75/d should be prescribed within 12 months.

SUMMARY:
The aim is to compare the results of using T-provisional and Mini-Crush stenting techniques in patients with bifurcation lesions in the CTO segment.

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for coronary angioplasty with stenting due to Ischemic heart disease (Stable angina, Unstable angina, non-ST Myocardial Infarction).
* Bifurcation side branch diameter >2 mm in CTO segment, verified by coronary angiography
* Successful CTO recanalization
* Signed, documented informed consent prior to admission to the study

Exclusion Criteria:

* Age <18 years or >75 years
* Left main artery bifurcation lesion
* Reocclusion CTOs
* Renal insufficiency (GFR/MDRD <30 ml/min)
* Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
* Known non-adherence to double anti-platelet therapy (DAPT)
* LVEF <30%
* Continuing bleeding
* Acute coronary syndrome (ST-elevation Myocardial infarction)
* Anamnesis of previous CABG
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | During 1 year after procedure
  Primary outcome is defined as a composite endpoint of cardiac death, target vessel myocardial infarction and clinically indicated target lesion revascularization.

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | During 1 year after procedure
  Major adverse cardiac and cerebrovascular events (MACCE) including: including: All-cause mortality, Myocardial infarction, Stent thrombosis, Clinically indicated Target lesion revascularization, Any target lesion revascularization, Any target vessel revascularization.
Restenosis of main vessel/side branch | At 12-month follow-up
  Angiographically estimated main vessel/side branch restenosis. Restenosis is defined as ≥ 50% diameter lumen loss in a target lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia